CLINICAL TRIAL: NCT05131334
Title: Auricular Vagus Nerve Stimulation (auriStim) Against Alcohol-craving Measured by Pupillary Reaction - Pilotstudy
Brief Title: Auricular Vagal Stimulation in Alcohol Craving
Acronym: VNS_CRAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Treiber, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2284/2017
Record Dates: First submitted 2021-10-15; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Alcohol Withdrawal; Psychophysiologic Reaction
Keywords: alcohol withdrawal; vagal stimulation; pupillometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Other): The pilot study applied an open-label, unblinded, repeated measures design with three time points of pupillometry measurements at two testing days. Patient serving as their own controls
  Interventions: Device: auriStim, for auricular vagal stimulation

INTERVENTIONS:
Device: auriStim, for auricular vagal stimulation — For auricular vagal stimulation we used auriStim (AU0115, Multisana GmbH, Vienna, Austria). Using a green light-emitting diode (LEDs) flashlight, blood vessels in the cymba conchae of the left ear side were detected. Minimal invasive needles (penetrating 1-2mm) were placed close to the vessel-bifurcation to provide efficient stimulation of the auricular branch of the vagus nerve. The built-in microchip controls monophasic volt pulses of 1 ms, with alternating polarity, a frequency of 1 Hz and an amplitude of 4V. Stimulation lasted for 72h in total with alternating on/off periods of three hours. Thereafter, the device was removed, and patients continued their therapy consisting of anti-withdrawal medication.

SUMMARY:
Background: The cause of the vegetative symptoms is a sympathetic driven misbalance of the autonomous nervous system. To restore vegetative balance in alcohol withdrawal syndrome new neuro-modulatory methods, such as percutaneous auricular vagal stimulation (pVNS) could be used. Measuring the pupil size is a suitable method to assess imbalances or dysfunctions of the vegetative regulation in individuals. Objective: The objective of this study is to assess the pupil reaction to the cholinergic antagonist tropicamide in alcohol withdrawal syndrome as a biomarker of the vegetative balance before and after pVNS. Methods: 30 patients aged between 20 and 65 were recruited in this open-label, controlled pilot trial with repeated measure design. pVNS was administered at the left cymba conchae for 72 hours with intermitted stimulation. Pupillometric recording lasted about 60 min and was performed at baseline and following pVNS. The reaction of the pupil to an anticholinergic agent was measured as a receptor-test in terms of a psychophysiological feedback mechanism to pVNS.

DETAILED DESCRIPTION:
The chronic consumption of alcohol leads to a pathophysiological adaptation of the nervous system, by an increase in glutamatergic receptors and a decrease in GABAergic receptor functions. Autonomic and psychomotor hyperactive disorders, such as nausea, tremor, diaphoresis, hypersensitive reflexes, hypertension, and tachycardia, as well as negative emotional states, characterized by restlessness, anxiety, dysphoria, and irritability occur 6 to 24 hours after cessation of alcohol consumption. The cause of the vegetative symptoms is a sympathetic driven misbalance of the autonomous nervous system. The negative state of health can last for a very long time and is the main reason for relapses.

Pharmacological treatment of alcohol withdrawal syndrome consists of ether Benzodiazepines or GHB is an endogenous metabolite of γ-aminobutyric acid (GABA).

The rate of successful treatment is lowest for alcohol dependence among all psychiatric disorders. Therefore, it seems important to carry out further interdisciplinary investigations in the direction of new and effective treatment methods. To restore vegetative balance in alcohol-withdrawal syndrome novel neuromodulatory approaches, such percutaneous auricular vagal stimulation (pVNS) could be beneficial.

The pupil size changes, like other physiological markers, e.g., hyperventilation, blood pressure and heart rate, serves as psychophysiological marker of the autonomic nervous system (ANS). Beside the fact that pupil size is determined by balance between the parasympathetic ANS (PANS) and the sympathetic ANS (SANS), measuring the static and dynamic pupillary diameters are suitable parameters measuring imbalances or dysfunction of the vegetative regulation. The pupil diameter oscillates spontaneously at low frequencies, which is an almost constant oscillatory change in the pupil size. Like pupil size, it is generally assumed that pupil oscillation is regulated by a dynamic interaction between parasympathetic (cholinergic) and sympathetic (noradrenergic) activity.

In this study, the investigator assessed the pupil reaction to the cholinergic antagonist tropicamide in alcohol withdrawal syndrome as a biomarker of the vegetative balance before and after pVNS. The Investigator hypothesized that pVNS will enhance the parasympathomimetic tone represented by a reduction of pupillary diameter in a parasympatholytic pharmacological challenge with tropicamide after vagal stimulation.

Study Design

The pilot study applied an open-label, unblinded, repeated measures design with three time points of pupillometry measurements at two testing days. For baseline measurements, the static pupil measurement was taken with the head fixed in a position and with open eyes (0'). Followed by an administration one drop of 0.01% tropicamide-solution into the left eye. The dynamic pupil measure followed 20 minutes (20') and 40 minutes (40') after tropicamide application. In our protocol the investigator scheduled a 60' measurement, which was removed due to the finding, that a maximum dilation was measured after 40' and that patients became increasingly agitated and weary, often leading to biased recordings at baseline measurement. Absolute change (mm), and relative change (%) of the pupil diameter was calculated.

Next, auriStim (AU0115, Multisana GmbH, Vienna, Austria) was placed for percutaneous vagal stimulation (pVNS). Patients were stimulated for 72 hours, with an intermittent stimulation mode, switching from active to resting state all three hours. After the stimulation period, patients placed their head in a fixed position for the second pupil measurement. For dynamic measurements, tropicamide was induced and measures were taken after 20' and 40'. Again, the investigator calculated absolute and relative changes of the pupil diameter. For each recording the investigator analyzed pupillary oscillations with a Fourier analysis as biomarker of the central nervous activation. All patients were tested at the same time of the day (between 9:00 and 10:00 a.m.) to exclude diurnal variation in pupillary diameter at day two and day five of the inpatient alcohol withdrawal.

Percutaneous auricular vagal nerve stimulation (pVNS)

For auricular vagal stimulation the investigator used auriStim (AU0115, Multisana GmbH, Vienna, Austria). Using a green light-emitting diode (LEDs) flashlight, blood vessels in the cymba conchae of the left ear side were detected. Minimal invasive needles (penetrating 1-2mm) were placed close to the vessel-bifurcation to provide efficient stimulation of the auricular branch of the vagus nerve. The built-in microchip controls monophasic volt pulses of 1 ms, with alternating polarity, a frequency of 1 Hz and an amplitude of 4V. Stimulation lasted for 72h in total with alternating on/off periods of three hours. Thereafter, the device was removed, and patients continued their therapy consisting of anti-withdrawal medication.

Quantitative pupillometry

Before recording, patients were acquainted to the test environment (160 lux) in a noise-protected room (3 x 4 meters) for three minutes. With head held steady in a chin- and forehead rest, the patients positioned their left eye in front of the camera and fixed a black dot, at 1.6m distance, to prevent accommodation. Pupillometry was performed using a non-invasive, personal computer-based infrared digital video pupillometer system (TV pupillometer 1050, Whittaker Corporation., California, Los Angeles). Incorporated five milliwatts, infra-red LEDs provide continuous illumination of the eye, with a wavelength of 850nm to achieve high contrast filming condition, and to which the pupil does not respond. The system integrates a calibrated light stimulation of fixed intensity (145 lux) and duration (300ms) to induce a light-evoked pupillary reaction. The system allows a precise (0.01mm limit) and rapid (50Hz) measure of the vertical diameter, and automatically determines static pupil size (averaged over the first 25.6sec of recording) and a series of dynamic pupillary parameters after light stimulation. Dynamic parameters include resting pupil diameter (pupil diameter just before light-stimulation), the latency for constriction (the latency time from the light flash exposure to the start of pupillary constriction), the amplitude of constriction (the value of the resting diameter minus the maximum constriction diameter), the constrictive ratio (amplitude of constriction/resting pupil diameter), the duration of constriction (time interval between the start of constriction, and the time point of maximum constriction) and peak constriction velocity. The recording of the pupillary diameter and response curve is shown as a graph of the pupillary diameter against time. Based on the measurement of static pupillary diameter (first 25.6sec) the pupillometer calculates pupillary oscillations by Fourier analysis (FA), reflecting the activation of the central nervous system. Prior to Fourier Analysis a linear interpolation was applied to artefacts such as blinking and missing data by a built-in noise removal program. For FA the investigator used five individual frequency bands: 0.0 - 0.2, 0.21 - 0.4, 0.41 - 0-6, 0.61 - 0.8, 0.81 - 1 Hz and whole power spectrum 0.0 - 1 Hz.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of alcohol dependence according to ICD-10 and DSM-V
* aged between 20 and 65
* Ability to perform oral and written informed consent to the study protocol

Exclusion Criteria:

* age under 20 or over 65 years
* taking medication affecting the pupillary measurements (opioids, acetylcholinesterase inhibitors, sympathomimetics)
* positive pregnancy test
* diagnosed anxiety disorders
* multiple substance abuse disorder
* ocular disease
* delirious patients
* biochemical implants
* hemophilia
* psoriasis vulgaris

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
mean pupillary diameter | 3 days
  change of the mean pupillary diameter in millimeter (mm), provoked by the parasympatholytic agent tropicamide (1 drop of 0.01% tropicamide solution administered into the left eye)

SECONDARY OUTCOMES:
resting pupillary diameter (millimeter) | 3 days
  pupil diameter just before light-stimulation
latency (milliseconds) | 3 days
  the latency time from the light flash exposure to the start of pupillary constriction
amplitude of constriction (millimeter) | 3 days
  the value of the resting diameter minus the maximum constriction diameter
constrictive ratio (percent) | 3 days
  amplitude of constriction/resting pupil diameter
duration of constriction (milliseconds) | 3 days
  time interval between the start of constriction, and the time point of maximum constriction
Pupillary oscillations (Hz) | 3 days
  Calculation of the pupillary oscillations by Fourier analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Henriette Walter, Prof., Principal Investigator — Department of Psychiatry and Psychotherapy, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Psychiatry and Psychotherapy, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No